CLINICAL TRIAL: NCT06833645
Title: To Investigate the Mechanism of Novel Molecular Probe [18F]AV45(Aβ) and [18F]AV1451(Tau)PET/CT in the Diagnosis of Early Pathological Changes of Alzheimer's Disease。
Brief Title: [18F]AV45(Aβ) and [18F]AV1451(Tau)PET/CT in the Diagnosis of Early Pathological Changes of Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Principal Investigator, Sichuan Provincial People's Hospital
Other Study IDs: SichuanPPH-AD
Record Dates: First submitted 2024-07-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Molecular Probes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild cognitive impairment，MCI
  Interventions: Other: molecular probe [18F]AV45(Aβ) and [18F]AV1451(Tau)
- Alzheimer's disease，AD
  Interventions: Other: molecular probe [18F]AV45(Aβ) and [18F]AV1451(Tau)
- Healthy volunteer
  Interventions: Other: molecular probe [18F]AV45(Aβ) and [18F]AV1451(Tau)

INTERVENTIONS:
Other: molecular probe [18F]AV45(Aβ) and [18F]AV1451(Tau) — The new imaging agents Aβ and TauPET/CT are molecular imaging, which have the advantage of earlier and more visual, and can study the mechanism of pathological changes and PET manifestations of Alzheimer's disease before symptoms appear from the molecular level.

SUMMARY:
To investigate the primary brain regions of precursors of Alzheimer's disease and Alzheimer's disease by novel molecular probe [18F]AV45(Aβ) and [18F]AV1451(Tau)PET/CT imaging. And the distribution of positive lesions in the brain area affecting the simple mental state examination and the Montreal Cognitive Assessment Scale in AD patients; It is expected to provide molecular imaging information for further study of the pathogenesis of AD. After clinical transformation, objective and quantitative positive diagnostic criteria for [18F]AV45 and [18F]AV1451PET/CT in the diagnosis of early Alzheimer's disease were established to avoid the defects of relying on the subjective experience of doctors and time-consuming diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Meet the MCI diagnostic criteria of Peterson in 2004;
* The clinicaldementiarating Scale (CDR) score was 0.5;
* Prominent memory loss may also be accompanied by impairment of other cognitive domains;
* Insidious onset and slow progression;
* Not at the level of dementia.

AD entry criteria:

* Meet the criteria for diagnosing dementia as described in the fourth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-R), Use the diagnostic criteria for AD from the National Institute of Neurology, Speech and Communication Disorders and Stroke - Alzheimer's Disease and Related Disorders (NINCDS-ADRDA) or the National Institute on Aging and Alzheimer's Disease Association (NIA-AA).
* Clinical Dementia Rating Scale score was 1 point.

Exclusion Criteria:

* Patients with a history of stroke and focal neurological signs, and imaging findings consistent with small cerebral vascular disease (Fazekas score ≥2);
* The presence of other neurological disorders that can cause brain dysfunction (e.g., depression, brain tumors, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, Normal facial pressure hydrocephalus);
* The presence of other systemic diseases that can cause cognitive impairment (such as liver insufficiency, renal insufficiency, thyroid dysfunction, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.);
* There is mental and neurological retardation.
* There are other diseases that are known to cause cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is expected to include 100 patients with MCI, 100 patients with AD, and 80 patients in the NC group, A total of 280 patients, all of whom received Aβ and TauPET/CT imaging. There were 180 males and 100 females.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-02-19 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
To establish diagnostic criteria of Aβ and TauPET/CT imaging | 2 months
  The areas of aβ and Tau positive lesions correlated with MMSE and MOCA scores were obtained.The SUVR cut-off values of aβ and Tau PET/CT for detecting positive lesions were obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Wang, Study Director — Sichuan Provincial People's Hospital
Locations (1):
- Departments of Nuclear Medicine, Sichuan Provincial People's Hospital, Chengdu, Sichuan, China